CLINICAL TRIAL: NCT03605056
Title: Chindamide in Combination With Lenalidomide and Dexamethasone for the Treatment of Relapsed/Refractory Multiple Myeloma, a Phase II Trial
Brief Title: Phase 2 Trial of Chidamide-Lenalidomide-Dexamethasone(CRD) Regimen in R/R MM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peng Liu (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Peng Liu, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHZS-MM001
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All the patients involved in this study will receive a 3-drug regimen (chindamide, lenalidomide and dexamethasone)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRD regimen (Experimental): CRD is a new 3-drug regimen adding a HDACi named chidamide to a novel 2-drug combination of lenalidomide and dexamethasone (RD)
  Interventions: Drug: chidamide; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: chidamide — 20 mg/d, will be administered orally, on Days 1, 4, 8, 11 of each 21 day cycle
  Other Names: Epidaza; CS055; HBI-8000
Drug: lenalidomide — 25 mg/d, will be administered orally on Days 1-14 each 21 day cycle
Drug: dexamethasone — 40mg weekly, will be administered orally or intravenously

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of combination of Chidamide-Lenalidomine-Dexamethasone in relapsed or refractory multiple myeloma patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ age 18 years
* Patient is able to understand and has given voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Patient has been previously diagnosed with MM based on standard International Myeloma Working Group (IMWG) criteria and currently requires treatment.
* Patient must have received at least one previous line of therapy for multiple myeloma including bortezomib
* Patient must have demonstrated disease progression on or within 60 days of completion of the last therapy. Patient has measurable disease defined as at least one of the following:
* Serum M protein ≥ 0.5 g/dL (≥5 g/L)
* Urine M protein ≥200 mg/24 hours
* Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Negative serum or urine pregnancy test for women of child-bearing potential
* Screening Laboratory parameters:
* Absolute neutrophil count (ANC) ≥ 1,500 cells/dL (1.5 x 10^9/L). Granulocyte colony-stimulating factor (GCSF) is not permitted during screening to meet eligibility criteria and within 14 days of initiation of therapy
* Platelet count ≥ 70,000 cells/dL (70 x 10^9/L) Platelet transfusion is not permitted during screening to meet eligibility criteria and within 14 days of initiation of therapy
* Hemoglobin ≥ 8.0 g/dl ( red blood cell (RBC) transfusions are permitted during the screening period)
* Total Bilirubin ≤ 1.5 X upper limit of normal (ULN) ; Aspartate transaminase (AST, or SGOT) and alanine transaminase (ALT, or SGPT) ≤ 2.5x ULN Estimated creatinine clearance by Cockcroft-Gault formula ≥ 50 mL/min

Exclusion Criteria:

* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy.
* Received any investigational drug within 14 days or 5 half-lives of the investigational drug, whichever is longer.
* Prior anti-cancer therapy within 14 days.
* Patient has any Grade 3 or > unresolved peripheral neuropathy from previous treatment.
* Patient is human immunodeficiency virus (HIV) positive,.
* Patient is Hepatitis B Surface antigen-positive or HBV-DNA copies > 10^3/ml
* Patient has active hepatitis C infection.
* Hypersensitivity to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs
* Known history of allergy to 2 or > drugs or any component of regimen
* Any clinically significant, uncontrolled medical conditions that, in the treating Investigator's opinion, would impose excessive risk to the patient or may interfere with compliance or interpretation of the study results. Uncontrolled intercurrent illness may include, but is not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations as determined by treating investigator that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-07-31 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 2 years
  according to IMWG criteria, including the rate of complete remission (CR), very good partial remission (VGPR) and partial remission (PR)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 2 years
  as assessed by CTCAE v4.0
Overall Survival Rate | 2 years
  The percentage of people in the study group who are still alive 2 years after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, MD,PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China